CLINICAL TRIAL: NCT04408157
Title: A Research Study to Evaluate the Efficacy of a Self-management Booklet (Stay Well During COVID-19; SWitCh) to Promote Wellbeing During the COVID-19 Pandemic
Brief Title: A Research Study to Evaluate the Benefits of a Self-management Booklet to Promote Wellbeing During the COVID-19 Pandemic
Acronym: SWitCh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: v1.1 06.05.2020
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2021-09

CONDITIONS: COVID
Keywords: wellbeing; covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Two-arm parallel randomised-controlled trial with nested qualitative study
Masking Description: Blinding not possible as passive control arm and using self-report outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-management booklet (Experimental): Self-management booklet: developed drawing on existing evidence and work conducted by researchers at the Health Psychology section at KCL, tailored to the current circumstances in response to the COVID-19 pandemic.
  Interventions: Behavioral: Self-management booklet (SWitCh: Stay well during COVID-19)
- Education only (waiting-list) (No Intervention): Participants allocated to the waiting-list control arm will receive a link via email to educational materials related to COVID produced by King's College London for an online event and will be provided with the self-management booklet after completing the T2 assessment and qualitative interview. The topics covered in the online event are the same as the ones included in the self-management booklet, without structured guidance and behaviour change techniques to facilitate behaviour change.

INTERVENTIONS:
Behavioral: Self-management booklet (SWitCh: Stay well during COVID-19) — The purpose of this booklet is to support adjustment to the current circumstances of the COVID-19 pandemic and facilitate the development and maintenance of healthy behaviours at home. The booklet covers a range of topics, including understanding bodily sensations and symptoms of COVID-19, managing the uncertainty surrounding COVID-19, physical activity, sedentary behaviour, sleep, social support and isolation, nutrition and alcohol consumption, sex and intimate relationships, and coping with children at home. The booklet will provide structured guidance on the various topics through the use of effective behaviour change techniques, in particular self-monitoring, goal setting, and problem solving and signposting to additional helpful resources, such as drinking or nutrition tracking apps.
  Arms: Self-management booklet

SUMMARY:
Background The immediate psychological impact of COVID-19 is already emerging. The investigators are interested in the benefits of a self-management booklet focused on the current circumstances in response to the COVID-19 pandemic on people's physical and mental wellbeing.

Who can participate? The investigators are looking for participants aged 18 and over who live in the UK and can read and write in English, without any current serious mental health problems (e.g. bipolar disorder, PTSD, active thoughts of self-harm, or severe anxiety/depression), and who feel that their physical and/or mental wellbeing have been affected since the COVID-19 pandemic.

What does the study involve? Eligible participants will complete questionnaires at baseline following which they will be randomly allocated to either receive the self-management booklet right away (via email) or after 4 months (waiting-list, in the meantime participants will be provided a link to educational materials). Participants will not be able to choose whether they will receive the self-management booklet right away or be in the waiting-list as a computer system (Qualtrics randomiser) will allocate them to one of the two groups at random. Participants in both conditions will be asked to complete online questionnaires at multiple time points, 2-months and 4-months after allocation. Participants in the waiting-list condition will also be asked to complete the same set of questionnaires at 6- and 8-months after allocation to assess how beneficial they found the self-management booklet.

Participants will also be invited to take part in an audio-recorded interview after T2 to tell us more about how they found the self-management booklet or the educational materials. The investigators will select 30 participants (15 from each condition) for the interview out of those who opt-in to capture a wide range of experiences and backgrounds.

What are the possible benefits and risks of participating? Risks to participants are small. Participants may find reflecting on the impact of COVID-19 on their lives distressing. However, these effects are anticipated to be short lived, as participants will learn psychological techniques during the intervention that can help them manage better in the current circumstances and improve their wellbeing.

Where is the study run from? The lead site is King's College London. The study is run online via Qualtrics.

When is the study starting and how long is it expected to run for? May 2020 to May 2021

Who is the main contact? Dr Federica Picariello federica.picariello@kcl.ac.uk

DETAILED DESCRIPTION:
In the UK, over 4 in 5 Britons are worried about the effect COVID-19 is having on their life, with over half reporting that their wellbeing has been affected. Providing support for individuals to build optimal structures to maintain their physical and mental wellbeing is key to mitigate the consequences of the pandemic on day-to-day life and in the longer term. The investigators would like to conduct a randomised-controlled trial to test the efficacy of a theory-based self-management booklet to improve physical and mental wellbeing versus education alone. The trial will include a nested qualitative study to explore in a subgroup of participants their experiences of the self-management booklet or education alone. The primary objective is to examine the efficacy of the self-management booklet at improving wellbeing as compared to the waiting-list control arm 2-months post-randomisation. The investigators also want to explore the treatment effects of the self-management booklet on secondary outcomes (health status, day-to-day activities, resilience, intolerance of uncertainty, loneliness, social support, sleep quality, napping, sedentary behaviour, physical activity, and COVID-19-related behaviours, symptom complaints). Tertiary objectives include exploring changes in self-reported primary and secondary outcomes over time in a non-randomised analysis combining data from both arms and qualitatively exploring participants' perceptions of the acceptability and usefulness of the self-management booklet. These objectives will be addressed by a two-armed parallel randomised controlled trial (RCT) with a nested qualitative study. The study will be conducted through Qualitrics (including recruitment, randomisation, and data collection). Participants in both arms will be followed-up at 2 and 4 months post-randomisation. Additionally, participants in the control arm will receive the self-management booklet after the 4-months follow-up assessment and will be followed-up at 6 and 8 months post-randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over who live in the UK and can read and write in English, without any current serious mental health problems (e.g. bipolar disorder, PTSD, active thoughts of self-harm, or severe anxiety/depression) and who feel that their physical and/or mental wellbeing have been affected since the COVID-19 pandemic.

Exclusion Criteria:

* Any current serious mental health problems (e.g. bipolar disorder, PTSD, active thoughts of self-harm, or severe anxiety/depression) or who feel that their physical and/or mental wellbeing have not been affected by COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS): Tennant et al., 2007 | 2 months post-randomisation
  validated self-report measure; scores range from 14 to 70 and higher scores indicate greater positive mental wellbeing.

SECONDARY OUTCOMES:
Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS): Tennant et al., 2007 | 4 months post-randomisation
  validated self-report measure; scores range from 14 to 70 and higher scores indicate greater positive mental wellbeing.
Self-rated health status: Bombak, 2013 | 2 months post-randomisation
  validated self-report measure; scores range from 0 to 100 and higher scores indicate better health
Self-rated health status: Bombak, 2013 | 4 months post-randomisation
  validated self-report measure; scores range from 0 to 100 and higher scores indicate better health
Brief Resilience Scale (BRS): Smith et al., 2008 | 2 months post-randomisation
  validated self-report measure; items are averaged to create a total score, ranging from 1 to 7 and higher total scores indicate higher levels of resilience.
Brief Resilience Scale (BRS): Smith et al., 2008 | 4 months post-randomisation
  validated self-report measure; items are averaged to create a total score, ranging from 1 to 7 and higher total scores indicate higher levels of resilience.
Intolerance of Uncertainty Scale (IUS-12): Carleton et al., 2007 | 2 months post-randomisation
  validated self-report measure; total scores range from 12 to 60 and higher scores indicate higher intolerance of uncertainty
Intolerance of Uncertainty Scale (IUS-12): Carleton et al., 2007 | 4 months post-randomisation
  validated self-report measure; total scores range from 12 to 60 and higher scores indicate higher intolerance of uncertainty
Positive Affect subscale of the Positive and Negative Affect Scale-X (PANAS-X): Watson & Clark, 1999 | 2 months post-randomisation
  validated self-report measure; positive affect items (N=27) are rated on a five-point scale (1) very slightly or not at all, (2) a little, (3) moderately, (4) quite a bit, and (5) extremely and can be grouped into subscales according to Watson, D., & Clark, L. A. (1999). The PANAS-X: Manual for the positive and negative affect schedule-expanded form. Higher scores indicate higher levels of positive affect states.
Positive Affect subscale of the Positive and Negative Affect Scale-X (PANAS-X): Watson & Clark, 1999 | 4 months post-randomisation
  validated self-report measure; positive affect items (N=27) are rated on a five-point scale (1) very slightly or not at all, (2) a little, (3) moderately, (4) quite a bit, and (5) extremely and can be grouped into subscales according to Watson, D., & Clark, L. A. (1999). The PANAS-X: Manual for the positive and negative affect schedule-expanded form. Higher scores indicate higher levels of positive affect states.
UCLA 3 item loneliness scale: Russell, 1996 | 2 months post-randomisation
  validated self-report measure; total scores range from 3 to 9 and higher scores indicate higher levels of loneliness
UCLA 3 item loneliness scale: Russell, 1996 | 4 months post-randomisation
  validated self-report measure; total scores range from 3 to 9 and higher scores indicate higher levels of loneliness
Multidimensional Scale of Perceived Social Support (MSPSS): Zimet et al., 1988 | 2 months post-randomisation
  validated self-report measure; the scale consists of three subscales (family, friends, and significant other) that contain 4 items each; each subscale score can range from 4 to 28. Items are summed, and a total score is also calculated and ranges from 12 to 84. Higher subscale and total scores indicate higher levels of perceived social support.
Multidimensional Scale of Perceived Social Support (MSPSS): Zimet et al., 1988 | 4 months post-randomisation
  validated self-report measure; the scale consists of three subscales (family, friends, and significant other) that contain 4 items each; each subscale score can range from 4 to 28. Items are summed, and a total score is also calculated and ranges from 12 to 84. Higher subscale and total scores indicate higher levels of perceived social support.
Subjective Health Complaint Scale (SHC): Eriksen, Ihlebæk, & Ursin, 1999 | 2 months post-randomisation
  validated self-report measure; a total score will be obtained for each symptom (severity x duration) with a possible range from 0 to 90, with higher scores indicating greater severity of a symptom, total number of symptoms reported, and a total score from 0 to 84 with higher scores indicating greater severity of somatic complaints.
Subjective Health Complaint Scale (SHC): Eriksen, Ihlebæk, & Ursin, 1999 | 4 months post-randomisation
  validated self-report measure; a total score will be obtained for each symptom (severity x duration) with a possible range from 0 to 90, with higher scores indicating greater severity of a symptom, total number of symptoms reported, and a total score from 0 to 84 with higher scores indicating greater severity of somatic complaints.
Leeds Sleep Evaluation Questionnaire (LSEQ): Parrott & Hindmarch, 1980 | 2 months post-randomisation
  validated self-report measure; responses are measured using a 100-mm scale and are then averaged to provide a score for each domain and higher scores indicate better sleep.
Leeds Sleep Evaluation Questionnaire (LSEQ): Parrott & Hindmarch, 1980 | 4 months post-randomisation
  validated self-report measure; responses are measured using a 100-mm scale and are then averaged to provide a score for each domain and higher scores indicate better sleep.
Self-reported napping: Stone et al., 2018 | 2 months post-randomisation
  self-report measure used in Stone et al., 2018; self-reported napping is defined as reporting at least 1 hour of napping each time and responses will be categorised as follows: no napping=coded as 0; <1 hour=coded as 1, 1-2 hours=coded as 2, and >2 hours=coded as 3.
Self-reported napping: Stone et al., 2018 | 4 months post-randomisation
  self-report measure used in Stone et al., 2018; self-reported napping is defined as reporting at least 1 hour of napping each time and responses will be categorised as follows: no napping=coded as 0; <1 hour=coded as 1, 1-2 hours=coded as 2, and >2 hours=coded as 3.
Work and Social Adjustment Scale (WSAS): Mundt et al., 2002 | 2 months post-randomisation
  validated self-report measure; total scores range from 0 to 40 and higher scores indicate greater impairment
Work and Social Adjustment Scale (WSAS): Mundt et al., 2002 | 4 months post-randomisation
  validated self-report measure; total scores range from 0 to 40 and higher scores indicate greater impairment
International Physical Activity Questionnaire -short form (IPAQ-SF): Craig et al., 2003 | 2 months post-randomisation
  validated self-report measure; The questionnaire can be scored categorically according to developed cut-offs to classify individuals into low, moderate, or high physical activity groups; or it can be scored continuously. Responses can be converted to Metabolic Equivalent Task minutes per week (METmin/wk), according to the IPAQ scoring protocol. MET scores across the three sub-components can be summed to indicate overall physical activity
International Physical Activity Questionnaire -short form (IPAQ-SF): Craig et al., 2003 | 4 months post-randomisation
  validated self-report measure; The questionnaire can be scored categorically according to developed cut-offs to classify individuals into low, moderate, or high physical activity groups; or it can be scored continuously. Responses can be converted to Metabolic Equivalent Task minutes per week (METmin/wk), according to the IPAQ scoring protocol. MET scores across the three sub-components can be summed to indicate overall physical activity

OTHER OUTCOMES:
COVID-related behaviours | Baseline (before randomisation), 2 and 4 months post-randomisation both arms, and 6 and 8 months post-randomisation control arm only.
  non-validated self-report items (such as following guidelines with regards to social distancing, rated from 0 to 10 with higher scores indicating better adherence to guidelines)
Change from baseline to follow-up on the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS): Tennant et al., 2007 | 4 months post-randomisbaseline (before randomisation), 2 and 4 months post-randomisation both arms, and 6 and 8 months post-randomisation control arm only (non-randomised comparison of change)
  validated self-report measure; scores range from 14 to 70 and higher scores indicate greater positive mental wellbeing.
Change from baseline to follow-up on the Self-rated health status: Bombak, 2013 | 4 months post-randomisbaseline (before randomisation), 2 and 4 months post-randomisation both arms, and 6 and 8 months post-randomisation control arm only (non-randomised comparison of change)
  validated self-report measure; scores range from 0 to 100 and higher scores indicate better health
Change from baseline to follow-up on the Brief Resilience Scale (BRS): Smith et al., 2008 | 4 months post-randomisbaseline (before randomisation), 2 and 4 months post-randomisation both arms, and 6 and 8 months post-randomisation control arm only (non-randomised comparison of change)
  validated self-report measure; items are averaged to create a total score, ranging from 1 to 7 and higher total scores indicate higher levels of resilience.
Change from baseline to follow-up on the Intolerance of Uncertainty Scale (IUS-12): Carleton et al., 2007 | 4 months post-randomisbaseline (before randomisation), 2 and 4 months post-randomisation both arms, and 6 and 8 months post-randomisation control arm only (non-randomised comparison of change)
  validated self-report measure; total scores range from 12 to 60 and higher scores indicate higher intolerance of uncertainty
Change from baseline to follow-up on the UCLA 3 item loneliness scale: Russell, 1996 | 4 months post-randomisbaseline (before randomisation), 2 and 4 months post-randomisation both arms, and 6 and 8 months post-randomisation control arm only (non-randomised comparison of change)
  validated self-report measure; total scores range from 3 to 9 and higher scores indicate higher levels of loneliness
Change from baseline to follow-up on the Multidimensional Scale of Perceived Social Support (MSPSS): Zimet et al., 1988 | 4 months post-randomisbaseline (before randomisation), 2 and 4 months post-randomisation both arms, and 6 and 8 months post-randomisation control arm only (non-randomised comparison of change)
  validated self-report measure; the scale consists of three subscales (family, friends, and significant other) that contain 4 items each; each subscale score can range from 4 to 28. Items are summed, and a total score is also calculated and ranges from 12 to 84. Higher subscale and total scores indicate higher levels of perceived social support.
Change from baseline to follow-up on the Leeds Sleep Evaluation Questionnaire (LSEQ): Parrott & Hindmarch, 1980 | 4 months post-randomisbaseline (before randomisation), 2 and 4 months post-randomisation both arms, and 6 and 8 months post-randomisation control arm only (non-randomised comparison of change)
  validated self-report measure; responses are measured using a 100-mm scale and are then averaged to provide a score for each domain and higher scores indicate better sleep.
Change from baseline to follow-up on the Work and Social Adjustment Scale (WSAS): Mundt et al., 2002 | 4 months post-randomisbaseline (before randomisation), 2 and 4 months post-randomisation both arms, and 6 and 8 months post-randomisation control arm only (non-randomised comparison of change)
  validated self-report measure; total scores range from 0 to 40 and higher scores indicate greater impairment
Change from baseline to follow-up on the International Physical Activity Questionnaire -short form (IPAQ-SF): Craig et al., 2003 | 4 months post-randomisbaseline (before randomisation), 2 and 4 months post-randomisation both arms, and 6 and 8 months post-randomisation control arm only (non-randomised comparison of change)
  validated self-report measure; The questionnaire can be scored categorically according to developed cut-offs to classify individuals into low, moderate, or high physical activity groups; or it can be scored continuously. Responses can be converted to Metabolic Equivalent Task minutes per week (METmin/wk), according to the IPAQ scoring protocol. MET scores across the three sub-components can be summed to indicate overall physical activity
Change from baseline to follow-up in self-reported napping: Stone et al., 2018 | 4 months post-randomisbaseline (before randomisation), 2 and 4 months post-randomisation both arms, and 6 and 8 months post-randomisation control arm only (non-randomised comparison of change)
  self-report measure used in Stone et al., 2018; self-reported napping is defined as reporting at least 1 hour of napping each time and responses will be categorised as follows: no napping=coded as 0; <1 hour=coded as 1, 1-2 hours=coded as 2, and >2 hours=coded as 3.
Change from baseline to follow-up on the Subjective Health Complaint Scale (SHC): Eriksen, Ihlebæk, & Ursin, 1999 | 4 months post-randomisbaseline (before randomisation), 2 and 4 months post-randomisation both arms, and 6 and 8 months post-randomisation control arm only (non-randomised comparison of change)
  validated self-report measure; a total score will be obtained for each symptom (severity x duration) with a possible range from 0 to 90, with higher scores indicating greater severity of a symptom, total number of symptoms reported, and a total score from 0 to 84 with higher scores indicating greater severity of somatic complaints.
Change from baseline to follow-up in Positive Affect states on the Positive and Negative Affect Scale-X (PANAS-X): Watson & Clark, 1999 | 4 months post-randomisbaseline (before randomisation), 2 and 4 months post-randomisation both arms, and 6 and 8 months post-randomisation control arm only (non-randomised comparison of change)
  validated self-report measure; positive affect items (N=27) are rated on a five-point scale (1) very slightly or not at all, (2) a little, (3) moderately, (4) quite a bit, and (5) extremely and can be grouped into subscales according to Watson, D., & Clark, L. A. (1999). The PANAS-X: Manual for the positive and negative affect schedule-expanded form. Higher scores indicate higher levels of positive affect states.

CONTACTS AND LOCATIONS:
Overall Officials: Federica Picariello, PhD, Principal Investigator — King's College London
Locations (1):
- Online recruitment through Qualtrics, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be confidentially and securely stored for 7 years as per University policy. Anonymised aggregated data will be made available upon request to the corresponding author.